CLINICAL TRIAL: NCT01515306
Title: A Study to Evaluate the Potential of Concomitant Ramucirumab to Affect the Pharmacokinetics of Paclitaxel in Patients With Advanced Malignant Solid Tumors
Brief Title: A Study of Ramucirumab (IMC-1121B) and Paclitaxel in Participants With Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14432; I4T-IE-JVCA (Other: Eli Lilly and Company); CP12-1032 (Other: ImClone Systems)
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Malignant Solid Tumor
Keywords: Advanced Malignant Solid Tumors
MeSH Terms: interventions — Ramucirumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A: ramucirumab (IMC-1121B) and paclitaxel (Experimental): Experimental: Part A: ramucirumab (IMC-1121B) and paclitaxel Cycle 1: paclitaxel administered on Day 1 of 2-week cycle. Cycle 2 and beyond : ramucirumab (IMC-1121B) administered on Day 1 and Day 15, paclitaxel administered on Day 1, Day 8 and Day 15 of 4-week cycle.
  Interventions: Biological: ramucirumab (IMC-1121B); Drug: paclitaxel
- Part B: ramucirumab (IMC-1121B) and paclitaxel (Experimental): Cycle 1: ramucirumab (IMC-1121B) administered as monotherapy on Day 1 of 3-week cycle.
  Cycle 2 and beyond: ramucirumab (IMC-1121B) administered on Day 1 and Day 15, paclitaxel administered on Day 1, Day 8 and Day 15 of 4- week cycle.
  *After Cycle 1 (mandatory pharmacokinetic phase) is completed, participants may continue to receive ramucirumab (IMC-1121B) monotherapy or combination therapy with paclitaxel as described in Part A.
  Interventions: Biological: ramucirumab (IMC-1121B); Drug: paclitaxel

INTERVENTIONS:
Biological: ramucirumab (IMC-1121B) — ramucirumab (IMC-1121B) 8 milligrams/kilogram (mg/kg) intravenous infusion, administered on Day 1and Day 15 of each 4-week cycle, unless otherwise specified.
  Other Names: LY3009806
Drug: paclitaxel — paclitaxel 80 milligrams/square meter (mg/m²) intravenous infusion, administered on Days 1, 8 and 15 of each 4-week cycle, unless otherwise specified.

SUMMARY:
The purpose of this study is to investigate whether there are no clinically significant pharmacokinetic effects of concomitant ramucirumab (IMC-1121B) on paclitaxel by investigating the pharmacokinetics (PK) of each in participants with advanced malignant solid tumors.

Part A of this study will investigate the potential of concomitant ramucirumab (IMC-1121B) to affect the pharmacokinetics of paclitaxel. Part B of this study will investigate the pharmacokinetics of ramucirumab (IMC-1121B) as monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Has histologic or cytologic documentation of a malignant solid tumor
* Has an advanced solid tumor that is refractory to standard therapy or for which no standard therapy is available
* Part A only: Has had 0-1 prior taxane-containing treatment regimens (including taxane monotherapy), which must have been completed at least 6 months before the first dose of study medication (prior bevacizumab is allowed)
* Part B only: Prior bevacizumab- and taxane-containing treatment regimens (including taxane monotherapy) are allowed, provided these regimens have been completed at least 6 months before the first dose of study medication
* Has resolution to Grade ≤ 1 of all clinically significant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy with the exception of peripheral neuropathy, which must not have exceeded Grade 1, by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI-CTCAE v 4.0)
* Has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 - 2
* Has adequate hematologic function. Blood transfusion is allowed but must be completed 48 hours before study drug administration
* Has adequate hepatic function (bilirubin ≤ 1.5 times the upper limit of normal [ULN], aspartate transaminase [AST] and alanine transaminase [ALT] ≤ 1.5 x ULN
* Has serum creatinine ≤ 1.5 x ULN. If serum creatinine > 1.5 x ULN, the calculated creatinine clearance (CrCl) should be ≥ 40 milliliter/minute (mL/min)
* Urinary protein is <2+ on dipstick or routine urinalysis (UA)
* Must have adequate coagulation function as defined by an international normalized ratio (INR) of ≤ 1.5 and a partial thromboplastin time (PTT) or an activated PTT (aPTT) ≤ 1.5 x ULN
* Eligible participants of reproductive potential agree to use adequate method of contraception during the study period and for 12 weeks after the last dose of study medication

Exclusion Criteria:

* Is receiving concomitant therapy with clinically relevant inhibitors or inducers of cytochrome P450, CYP2C8, CYP3AY and/or isoenzymes
* Are currently enrolled in, or discontinued within the last 14 days from, a clinical trial involving an investigational product or non-approved use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Has received a monoclonal antibody within 42 days prior to first dose of study medication
* Has received radiotherapy within 14 days prior to first dose of study medication
* Has received cytotoxic chemotherapy within 21 days (6 weeks for nitrosoureas or mitomycin C) prior to first dose of study medication
* Has a cardiac left ventricular ejection fraction (LVEF) not within institutional limits of normal on a multigated acquisition scan (MUGA) or echocardiogram
* Is receiving concurrent treatment with another anticancer therapy, including chemotherapy, immunotherapy, hormonal therapy, radiation therapy, chemoembolization, targeted or other investigational anticancer therapy
* Is receiving chronic therapy with nonsteroidal anti-inflammatory agents or other antiplatelet agents. Aspirin use at doses up to 325 milligrams/day (mg/day) and analgesic agents with no or low bleeding risk are permitted
* Has a history of uncontrolled hereditary or acquired bleeding or thromboembolic disorders
* Has experienced any arterial thromboembolic event, including myocardial infarction (MI), unstable angina stroke or transient ischemic attack (TIA), within 6 months prior to first dose of study medication
* Has a history of deep vein thrombosis, pulmonary embolism, or any other significant thromboembolism during the 3 months prior to first dose of study medication
* Has experienced a Grade 3 or 4 hemorrhagic event within 3 months prior to first dose of study medication
* Has experienced peripheral neuropathy ≥ Grade 2 at any time prior to study entry
* Has a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection, Crohn's disease, ulcerative colitis, or chronic diarrhea
* History of gastrointestinal perforation and / or fistulae within 6 months prior to randomization
* Has an ongoing or active infection requiring treatment with intravenous antibiotics
* Has a serious or nonhealing wound, peptic ulcer, or bone fracture within 28 days prior to first dose of study medication
* Has uncontrolled hypertension
* Has symptomatic congestive heart failure
* Has known brain or leptomeningeal disease
* Has known positive status for human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome-related illness
* Has known active drug or alcohol abuse that would affect participant's ability to comply with study treatment
* Has pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen
* Has had major surgery within 28 days prior to first dose of study medication or subcutaneous venous access device implantation within 7 days prior to first dose of study medication
* Has an elective or planned major surgery during the course of the trial
* If a primary cancer is non-small-cell lung cancer (NSCLC), participant has intratumor cavitation, radiologically documented evidence of major blood vessel invasion or encasement by cancer, or proximity of cancer to major airways
* Has received prior ramucirumab (IMC-1121B) therapy
* The participant has:

  * cirrhosis at a level of Child-Pugh B (or worse)
  * cirrhosis (any degree) and a history of hepatic encephalopathy or ascites resulting from cirrhosis and requiring ongoing treatment with diuretics and/or paracentesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-07-19 (Actual); Primary Completion 2013-03-20 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (6):
  - ImClone Investigational Site, Ann Arbor, Michigan
  - ImClone Investigational Site, Detroit, Michigan
  - ImClone Investigational Site, New Brunswick, New Jersey
  - ImClone Investigational Site, Cleveland, Ohio
  - ImClone Investigational Site, Philadelphia, Pennsylvania
  - ImClone Investigational Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Paclitaxel and Ramucirumab: Cycle 1: paclitaxel 80 milligrams/square meter (mg/m²) administered on Day 1 of 2-week cycle.
  Cycle 2 and beyond: ramucirumab (IMC-1121B) 8 milligrams/kilogram (mg/kg) administered on Day 1 and Day 15, paclitaxel 80 mg/m² administered on Day 1, Day 8 and Day 15 of 4-week cycle.
- Part B: Ramucirumab With or Without Paclitaxel: Cycle 1: ramucirumab (IMC-1121B) 8 mg/kg administered as monotherapy on Day 1 of 3-week cycle.
  Cycle 2 and beyond: ramucirumab (IMC-1121B) 8 mg/kg administered on Day 1 and Day 15, paclitaxel 80 mg/m² administered on Day 1, Day 8 and Day 15 of 4-week cycle.
  *After Cycle 1 (mandatory pharmacokinetic phase) is completed, participants may continue to receive ramucirumab (IMC-1121B) monotherapy or combination therapy with paclitaxel as described in Part A.
Period: Overall Study
Arm/Group | Part A: Paclitaxel and Ramucirumab | Part B: Ramucirumab With or Without Paclitaxel
Started | 24 | 16
Received at Least 1 Dose of Study Drug | 24 | 16
Cycle 1 | 24 | 16
Cycle 2 | 21 | 15
Drug-Drug Interaction Population | 21 (Completed Cycle 1 Day 1 and Cycle 2 Day 1 treatment.) | 0 (Drug-drug interaction was only assessed in Part A.)
Completed | 0 | 2
Not Completed | 24 | 14
Not completed — Adverse Event | 3 | 2
Not completed — Progressive Disease | 19 | 9
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Paclitaxel and Ramucirumab | Part B: Ramucirumab With or Without Paclitaxel | Total
Number analyzed (Participants) | 24 | 16 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 10 | 24
  >=65 years | 10 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 11 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 23 | 16 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 15 | 37
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 16 | 40

OUTCOME MEASURES:

1. Primary Outcome: Part A: Pharmacokinetics - Dose-Normalized Area Under the Concentration Versus Time Curve of Paclitaxel From Time Zero to Infinity [AUC(0-∞)] in Cycle 1
Description: Dose-normalized AUC(0-∞) was calculated from AUC(0-∞) divided by the dose. Data presented are Geometric Least Squares (Geo LS) means. Geo LS means were adjusted for cycle, participant and random error.
Time Frame: Cycle 1: 0, 1, 1.5, 2, 5, 7, 24, 48, 72 and 168 hours post paclitaxel infusion
Population: All participants from Part A Cycle 1 and had sufficient concentration data to calculate paclitaxel AUC(0-∞).
Measure: Least Squares Mean (90% Confidence Interval); unit: nanograms*hour/milliliter/milligram
Groups:
- Part A: Paclitaxel Alone (Cycle 1): Cycle 1: paclitaxel 80 milligrams/square meter (mg/m²) administered on Day 1 of 2-week cycle.
Arm/Group | Part A: Paclitaxel Alone (Cycle 1)
Number analyzed (Participants) | 19
nanograms*hour/milliliter/milligram | 29 [24.50 to 34.34]

2. Primary Outcome: Part A: Pharmacokinetics - Dose-Normalized Area Under the Concentration Versus Time Curve of Paclitaxel From Time Zero to Infinity [AUC(0-∞)] in Cycle 2
Description: as for outcome 1
Time Frame: Cycle 2: -1, 0, 1, 1.5, 2, 5, 7, 24, 48, 72, 96, 168, 264 and 336 hours post paclitaxel infusion
Population: All participants from Part A Cycle 2 and had sufficient concentration data to calculate paclitaxel AUC(0-∞).
Measure: Least Squares Mean (90% Confidence Interval); unit: nanograms*hour/milliliter/milligram
Groups:
- Part A: Paclitaxel + Ramucirumab (Cycle 2): Cycle 2: ramucirumab (IMC-1121B) 8 milligrams/kilogram (mg/kg) administered on Day 1 and Day 15, paclitaxel 80 mg/m² administered on Day 1, Day 8 and Day 15 of 4-week cycle.
Arm/Group | Part A: Paclitaxel + Ramucirumab (Cycle 2)
Number analyzed (Participants) | 17
nanograms*hour/milliliter/milligram | 31.67 [26.58 to 37.73]
Statistical Analysis 1: Comparison: Part A: Paclitaxel + Ramucirumab (Cycle 2); Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geo LS mean is AUC(0-∞) of Cycle 2/Cycle 1; Ratio of Geo LS means = 1.09, 90% CI 2-sided [0.93 to 1.29]

3. Primary Outcome: Part A: Pharmacokinetics - Dose-Normalized Maximum Observed Drug Concentration (Cmax) of Paclitaxel in Cycle 1
Description: Dose-normalized Cmax was calculated from Cmax divided by the dose. Data presented are Geometric Least Squares (Geo LS) means. Geo LS means were adjusted for cycle, participant and random error.
Time Frame: Cycle 1: 0,1, 1.5, 2, 5, 7, 24, 48, 72 and 168 hours post paclitaxel infusion
Population: All participants from Part A Cycle 1 and had sufficient concentration data to calculate paclitaxel cmax.
Measure: Least Squares Mean (90% Confidence Interval); unit: nanograms/milliliter/milligram
Arm/Group | Part A: Paclitaxel Alone (Cycle 1)
Number analyzed (Participants) | 21
nanograms/milliliter/milligram | 18.84 [16.03 to 22.13]

4. Primary Outcome: Part A: Pharmacokinetics - Dose-Normalized Maximum Observed Drug Concentration (Cmax) of Paclitaxel in Cycle 2
Description: as for outcome 3
Time Frame: Cycle 2: -1, 0, 1, 1.5, 2, 5, 7, 24, 48, 72, 96, 168, 264 and 336 hours post paclitaxel infusion
Population: All participants from Part A Cycle 2 and had sufficient concentration data to calculate paclitaxel cmax.
Measure: Least Squares Mean (90% Confidence Interval); unit: nanograms/milliliter/milligram
Arm/Group | Part A: Paclitaxel + Ramucirumab (Cycle 2)
Number analyzed (Participants) | 20
nanograms/milliliter/milligram | 18.30 [15.54 to 21.56]
Statistical Analysis 1: Comparison: Part A: Paclitaxel + Ramucirumab (Cycle 2); Test type: Superiority or Other; Mixed Models Analysis; Ratio of Geo LS mean is Cmax of Cycle 2/Cycle 1; Ratio of Geo LS means = 0.97, 90% CI 2-sided [0.83 to 1.13]

5. Primary Outcome: Part B: Pharmacokinetics - Dose-Normalized Area Under the Concentration Versus Time Curve of Ramucirumab From Time Zero to Infinity [AUC(0-∞)] as Monotherapy
Description: Dose-normalized AUC(0-∞) was calculated from AUC(0-∞) divided by the dose.
Time Frame: Cycle 1: 0,1, 1.5, 2, 5, 7, 24, 48, 72,168, 264, 336, 408, and 504 hours post ramucirumab infusion
Population: All participants who received ramucirumab and had sufficient concentration data to calculate ramucirumab AUC(0-∞) in Cycle 1 of Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliter/milligram
Groups:
- Part B: Ramucirumab Alone (Cycle 1): Cycle 1: ramucirumab (IMC-1121B) 8 mg/kg administered as monotherapy on Day 1 of 3-week cycle.
Arm/Group | Part B: Ramucirumab Alone (Cycle 1)
Number analyzed (Participants) | 15
micrograms*hour/milliliter/milligram | 55.3 (27)

6. Secondary Outcome: Part A: Pharmacokinetics - Dose-Normalized Area Under the Concentration Versus Time Curve of Ramucirumab From Time Zero to Infinity [AUC(0-∞)] in the Presence of Paclitaxel
Description: Dose-normalized AUC(0-∞) was calculated from AUC(0-∞) divided by the dose.
Time Frame: Cycle 2: 0, 1, 2, 2.5, 3, 6, 8, 25, 49, 73, 97, 169, 265 and 337 hours post ramucirumab infusion
Population: All participants who received ramucirumab and paclitaxel and had sufficient concentration data to calculate ramucirumab AUC(0-∞) in Cycle 2 of Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliters/milligram
Arm/Group | Part A: Paclitaxel + Ramucirumab (Cycle 2)
Number analyzed (Participants) | 13
micrograms*hour/milliliters/milligram | 55.4 (27)

7. Secondary Outcome: Part A: Pharmacokinetics - Dose-Normalized Maximum Observed Drug Concentration (Cmax) of Ramucirumab in the Presence of Paclitaxel
Description: Dose-normalized Cmax was calculated from Cmax divided by the dose.
Time Frame: Cycle 2: 0, 1, 2, 2.5, 3, 6, 8, 25, 49, 73, 97, 169, 265 and 337 hours post ramucirumab infusion
Population: All participants who received ramucirumab and paclitaxel and had sufficient concentration data to calculate ramucirumab Cmax in Cycle 2 of Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter/milligram
Arm/Group | Part A: Paclitaxel + Ramucirumab (Cycle 2)
Number analyzed (Participants) | 21
micrograms/milliliter/milligram | 0.384 (31)

8. Secondary Outcome: Part A: Immunogenicity of Ramucirumab in Combination With Paclitaxel - Number of Participants With Anti-Ramucirumab Antibodies
Description: Number of participants with positive treatment emergent anti-ramucirumab antibodies was summarized by treatment group. A treatment-emergent anti-drug antibodies (TEADA) sample was defined as: a post treatment sample with at least a 4-fold increase in titer from pre treatment sample; or 1:20 post treatment titer for participants that had no detectable ADA titer at baseline.
Time Frame: -1 hour on Day 1 of Cycle 2, and 30 days after last dose of study drug
Population: All participants from Part A Cycle 2, who received ramucirumab and paclitaxel and had data for anti-ramucirumab antibodies.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Paclitaxel and Ramucirumab (Cycle 2): Cycle 2: ramucirumab (IMC-1121B) 8 milligrams/kilogram (mg/kg) administered on Day 1 and Day 15, paclitaxel 80 mg/m² administered on Day 1, Day 8 and Day 15 of 4-week cycle.
Arm/Group | Part A: Paclitaxel and Ramucirumab (Cycle 2)
Number analyzed (Participants) | 10
Participants | 0

9. Secondary Outcome: Part B: Immunogenicity of Ramucirumab as Monotherapy - Number of Participants With Anti-Ramucirumab Antibodies
Description: as for outcome 8
Time Frame: 0 hour on Day 1 of Cycle 1, and 30 days after last dose of study drug
Population: All participants from Part B cycle 1, who received ramucirumab and had data for anti-ramucirumab antibodies.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Ramucirumab Alone (Cycle 1)
Number analyzed (Participants) | 1
Participants | 0

ADVERSE EVENTS:
Time Frame: Baseline, up to 8 years
Description: All participants who received at least one dose of study drug.
Groups:
- Part B: Ramucirumab + Paclitaxel (Cycle 2): Cycle 2 and beyond: ramucirumab (IMC-1121B) 8 mg/kg administered on Day 1 and Day 15, paclitaxel 80 mg/m² administered on Day 1, Day 8 and Day 15 of 4-week cycle.
Arm/Group | Part A: Paclitaxel Alone (Cycle 1) | Part A: Paclitaxel + Ramucirumab (Cycle 2) | Part B: Ramucirumab Alone (Cycle 1) | Part B: Ramucirumab + Paclitaxel (Cycle 2)
Serious Adverse Events (participants affected / at risk) | 1/24 | 6/21 | 0/16 | 6/15
Other Adverse Events (participants affected / at risk) | 18/24 | 21/21 | 8/16 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Paclitaxel Alone (Cycle 1) (N=24) | Part A: Paclitaxel + Ramucirumab (Cycle 2) (N=21) | Part B: Ramucirumab Alone (Cycle 1) (N=16) | Part B: Ramucirumab + Paclitaxel (Cycle 2) (N=15)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Paclitaxel Alone (Cycle 1) (N=24) | Part A: Paclitaxel + Ramucirumab (Cycle 2) (N=21) | Part B: Ramucirumab Alone (Cycle 1) (N=16) | Part B: Ramucirumab + Paclitaxel (Cycle 2) (N=15)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 10 (12) | 0 (0) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (10) | 0 (0) | 3 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (3)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Breath odour (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (3) | 1 (1) | 3 (3)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 8 (9) | 1 (1) | 3 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (9) | 4 (4) | 4 (4)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 4 (5) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (7) | 2 (2) | 2 (2)
Application site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 14 (17) | 2 (2) | 4 (6)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (3)
Oedema peripheral (General disorders) | 0 (0) | 5 (7) | 1 (1) | 4 (5)
Pyrexia (General disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Thrombosis in device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (6) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (5)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 3 (4) | 1 (1) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (5)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 6 (8) | 1 (1) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 7 (8) | 0 (0) | 2 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 4 (5) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3) | 4 (6)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 1 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7) | 0 (0) | 6 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (6) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 5 (6) | 1 (1) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.